CLINICAL TRIAL: NCT06516861
Title: Comparison of Magnesium Sulphate 30 mg/Kg With Lidocaine 1,5 mg/Kg in Hemodynamic Changes and Cortisol Level Post-intubation in Patient Undergoing Craniotomy
Brief Title: Magnesium Sulphate and Lidocaine in Hemodynamic Changes and Cortisol Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arsil Radiansyah (Other)
Collaborators: Universitas Sumatera Utara (Other)
Responsible Party: Sponsor-Investigator, Arsil Radiansyah, Resident Doctor, Universitas Sumatera Utara
Organization: Universitas Sumatera Utara (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: USumateraUtara01
Record Dates: First submitted 2024-06-23; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Intubation Complication
Keywords: Craniotomy; Intubation; Lidocaine; MgSO4
MeSH Terms: interventions — Magnesium Sulfate; Lidocaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: The design of this study used a double-blind randomized controlled clinical trial with pre test post test with control group design, to assess the comparison of hemodynamics and post-intubation cortisol in the administration of intravenous Magnesium sulfate and intravenous Lidocaine. The study sample was all patients who underwent surgery who met the inclusion and exclusion criteria.
Who Masked: Participant, Care Provider
Masking Description: masks the subjects and care provider from knowing which study treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MgSO4 intravenous (Experimental): Sample will be given MgSO4 30mg/Kg Intravenous as a premedication drugs before intubation for all patients who had craniotomy surgery
  Interventions: Drug: Magnesium Sulfate 20 MG/ML
- Lidocaine intravenous (Experimental): Sample will be given Lidocain 1.5mg/Kg Intravenous as a premedication drugs before intubation for all patients who had craniotomy surgery
  Interventions: Drug: Lidocaine IV
- NaCl 0,9% Intravenous (Placebo Comparator): Sample will be given NaCl 0,9% Intravenous 20 ml as a premedication drugs before intubation for all patients who had craniotomy surgery
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: Magnesium Sulfate 20 MG/ML — Administered intravenously with a dose of 30 mg/kg
  Other Names: Magnesium sulfate injection
  Arms: MgSO4 intravenous
Drug: Lidocaine IV — Administered intravenously with a dose of 1.5mg/Kg
  Other Names: Lidocaine
  Arms: Lidocaine intravenous
Drug: saline solution — Administered intravenously with 20 ml
  Other Names: NaCl 0,9% Solution
  Arms: NaCl 0,9% Intravenous

SUMMARY:
The sample was randomly divided into 3 groups consisting of patients who received Magnesium Sulfate 30 mg/Kg, Lidocaine 1.5 mg/Kg, and Control. These groups will be checked for hemodynamic changes and cortisol values.

DETAILED DESCRIPTION:
The sample was randomly divided into 3 groups and divided into 3 groups consisting of patients who received Magnesium Sulfate 30 mg/Kg, Lidocaine 1.5 mg/Kg, and Control. The first group of patients was given Magnesium Sulfate 30 mg /kg diluted in 20 ml with NaCl 0.9%, labeled with code A, and given in 5 minutes with a syringe pump, The second group was given Lidocaine 1.5 mg/kg diluted in 20 ml with NaCl 0.9%, labeled with code B and given in 5 minutes with a syringe pump, The third group was given NaCl 0.9%, in a 20 ml syringe labeled with code C and given in 5 minutes with a syringe pump. After induction and intubation, patients were then recorded systolic blood pressure, diastolic blood pressure, MAP, and pulse at T1 (3 minutes), T2 (5 minutes), T3 (7 minutes), and T4 (10 minutes).

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-65 years;
* body mass index (BMI) 18.5 kg/m2 - 29.9 kg/m2;
* patients or their families agreed to be used as research subjects;
* elective non-traumatic craniotomy cases, namely supratentorial brain tumor evacuation, intracerebral hemorrhage evacuation, subdural hemorrhage, cerebrovascular correction.

Exclusion Criteria:

* cardiac, hepatic, and renal disorders;
* patients with pregnancy;
* hypertension or hypotension before surgery;
* hypersensitivity to Magnesium Sulfate and/or Lidocaine;
* patients with chronic use of corticosteroid drugs, calcium channel blockers, magnesium-containing drugs, and opioids;
* risk of difficult intubation and ventilation according to the LEMON score and MOANS score criteria;
* impaired cortisol secretion (pituitary tumor or hypothalamic tumor or adrenal gland disorder); and
* patients with hypocortisol or hypercortisol at T0 serum cortisol examination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 1 month
  mmHg
Diastolic Blood Pressure | 1 month
  mmHg
Mean Arterial Pressure (MAP) | 1 month
  Estimated by using a formula in which the lower (diastolic) blood pressure is doubled and added to the higher (systolic) blood pressure and that composite sum then is divided by 3 to estimate MAP
Heart Rate | 1 month
  beats per minute

SECONDARY OUTCOMES:
Cortisol Levels | 1 month
  Cortisol Levels in nmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Rr Sinta Irina, MD, Study Chair — Universitas Sumatera Utara
Locations (1):
- Adam Malik General Hospital, Medan, North Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bousselmi R, Lebbi MA, Bargaoui A, Ben Romdhane M, Messaoudi A, Ben Gabsia A, Ferjani M. Lidocaine reduces endotracheal tube associated side effects when instilled over the glottis but not when used to inflate the cuff: A double blind, placebo-controlled, randomized trial. Tunis Med. 2014 Jan;92(1):29-33. PMID 24879167
- [Result] Silpa AR, Koshy KA, Subramanian A, Pradeep KK. Comparison of the efficacy of two doses of dexmedetomidine in attenuating the hemodynamic response to intubation in patients undergoing elective cardiac surgery: A randomized double-blinded study. J Anaesthesiol Clin Pharmacol. 2020 Jan-Mar;36(1):83-87. doi: 10.4103/joacp.JOACP_235_18. Epub 2020 Feb 18. PMID 32174664
- [Result] Sriganesh K, Syeda S, Shanthanna H, Venkataramaiah S, Palaniswamy SR. Effect of Opioid Versus Non-Opioid Analgesia on Surgical Pleth Index and Biomarkers of Surgical Stress During Neurosurgery for Brain Tumors: Preliminary Findings. Neurol India. 2020 Sep-Oct;68(5):1101-1105. doi: 10.4103/0028-3886.294559. PMID 33109859
- [Result] Finnerty CC, Mabvuure NT, Ali A, Kozar RA, Herndon DN. The surgically induced stress response. JPEN J Parenter Enteral Nutr. 2013 Sep;37(5 Suppl):21S-9S. doi: 10.1177/0148607113496117. PMID 24009246
- [Result] Rastogi, S., Yadav, S. K., Agarwal, A., Kumar, S., & Malviya, D. (2020). Biochemical markers and haemodynamic changes of stress response after intubation with direct laryngoscopy versus video laryngoscopy versus fiberoptic intubation: A comparative study. Indian Journal of Clinical Anaesthesia, 7(4), 681-686.
- [Result] Prete A, Yan Q, Al-Tarrah K, Akturk HK, Prokop LJ, Alahdab F, Foster MA, Lord JM, Karavitaki N, Wass JA, Murad MH, Arlt W, Bancos I. The cortisol stress response induced by surgery: A systematic review and meta-analysis. Clin Endocrinol (Oxf). 2018 Nov;89(5):554-567. doi: 10.1111/cen.13820. Epub 2018 Aug 23. PMID 30047158
- [Result] Gil-Gouveia R, Goadsby PJ. Neuropsychiatric side-effects of lidocaine: examples from the treatment of headache and a review. Cephalalgia. 2009 May;29(5):496-508. doi: 10.1111/j.1468-2982.2008.01800.x. Epub 2009 Feb 24. PMID 19250287
- [Result] Misganaw A, Sitote M, Jemal S, Melese E, Hune M, Seyoum F, Sema A, Bimrew D. Comparison of intravenous magnesium sulphate and lidocaine for attenuation of cardiovascular response to laryngoscopy and endotracheal intubation in elective surgical patients at Zewditu Memorial Hospital Addis Ababa, Ethiopia. PLoS One. 2021 Jun 1;16(6):e0252465. doi: 10.1371/journal.pone.0252465. eCollection 2021. PMID 34061894
- [Result] Mendonca FT, de Queiroz LM, Guimaraes CC, Xavier AC. Effects of lidocaine and magnesium sulfate in attenuating hemodynamic response to tracheal intubation: single-center, prospective, double-blind, randomized study. Braz J Anesthesiol. 2017 Jan-Feb;67(1):50-56. doi: 10.1016/j.bjane.2015.08.004. Epub 2016 Nov 22. PMID 28017170

DOCUMENTS (1):
  • Study Protocol (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT06516861/Prot_000.pdf